CLINICAL TRIAL: NCT03164174
Title: Atherosclerosis-Progression in Coronary Arteries Compared to Periphery Vessels
Acronym: APRICOTS
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Peter Marschang, Ao.Univ.Prof.Dr., Medical University Innsbruck
Other Study IDs: AN2016-0188 366/4.3
Record Dates: First submitted 2017-05-16; First posted 2017-05-23 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The study is a prospective-observational, explorative single-centre cohort study aimed to examine the atherosclerosis progression in coronary arteries compared to peripheral vessels (carotids, femoral arteries). Atherosclerotic alterations in peripheral vessels (IMT, plaque volume, plaque morphology) will be measured with ultrasound (IMT measurements and 3D quantitative plaque volumetry), whereas atherosclerotic alterations in coronary arteries will be tested with cardiac computertomography (CT) (coronary artery calcium score, calcium volume score, plaque morphology).

A total of 55 patients without prior known established vascular diseases will be tested. Cardiac CT and ultrasonography will be performed initially. After 2 years follow-up CT and ultrasound examination will be performed to assess the changes in atherosclerotic burden. Initially and after two years plasma samples will be collected and tested for traditional and novel cardiovascular risk factors.

The primary endpoint of the planned study will be the correlation of the atherosclerotic progression between coronary arteries and peripheral arteries (carotids, femoral arteries).

Secondary endpoints will include the correlation of atherosclerotic progression with established (hypertension, smoking, diabetes, dyslipidemia) and novel risk factors (hsCRP, P-selectin, cholesteryl ester transfer protein (CETP), intercellular adhesion molecule-1 (ICAM-1), CETP TaqIb polymorphism), with cardiovascular event rate, and the additional predictive value of atherosclerotic progression compared to an established risk score (SCORE Card, FRS). Also plaque morphology will be compared between coronary arteries and peripheral vessels.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-85 years, no prior established vascular diseases (CAD, PAD, cerebrovascular disease) no diabetes

Exclusion Criteria:

* Prior myocardial revascularisation therapy (aortocoronary bypass, PCI with stent implantation), coronary artery disease (CAD), peripheral artery disease (PAD), cerebrovascular disease (e.g.stroke), diabetes, pregnancy, lactation period, chronic renal insufficiency IIIB or lower (GFR <45ml/min), manifest hyperthyreosis

Ages: 30 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Non-diabetic patients without prior established vascular diseases (CAD, PAD, cerebrovascular disease) will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of the atherosclerotic progression between coronary arteries and peripheral arteries | 2 years
  Atherosclerotic progression in peripheral vessels (carotids, femoral arteries) will be tested with 3D-ultrasonography and a quantitative 3-D Plaque volumetry will be performed (total plaque volume).Atherosclerotic progression in coronary arteries will be measured with cardiac CT and coronary plaque burden will be assessed (calcium volume score). The percent change of atherosclerotic progression in peripheral vessels (percent change in total plaque volume, mm3) and coronary arteries (percent change in calcium score, Agatston units) will be compared.

SECONDARY OUTCOMES:
Correlation of atherosclerotic progression with established cardiovascular risk factors | 2 years
  Atherosclerotic Progression will be measured as stated above (total plaque volume for peripheral vessels, calcium volume score for coronary arteries). Cardiovascular risk factors include hypertension, smoking, diabetes, dyslipidemia
Correlation of atherosclerotic progression with novel cardiovascular risk factors | 2 years
  Atherosclerotic progression will be measured as stated above. Novel cardiovascular risk factors include hsCRP, P-selectin, cholesteryl ester transfer protein (CETP), intercellular adhesion molecule-1 (ICAM-1), CETP TaqIb polymorphism, lipocalin,catestatin.
Correlation of atherosclerotic progression with cardiovascular event rate | 2 years
  Atherosclerotic Progression will be measured as stated above. Cardiovascular event rate include MACCE (Major Adverse Cardiac and Cerebrovascular Events)
Additional predictive value of atherosclerotic progression compared to an established risk score (SCORE Card, FRS). | 2 years
  Atherosclerotic Progression will be measured as stated above. Established risk scores include SCORE and FRS.
Comparison of plaque morphology between coronary arteries and peripheral vessels | 2 years
  Plaque morphology in peripheral arteries will be measured with ultrasound. Therefore Gray-Weale-Score, Grey scale median and plaque structure will be assessed. For cardiac CT the noncalcifying burden atheroma score and high risk plaque criteria will be measured. Plaque morphology in peripheral arteries as measured by ultrasound and in coronary arteries as determined by CT will be compared in a qualitative manner.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria